CLINICAL TRIAL: NCT06115603
Title: CBG and Attention: A Double-Blind, Randomized, Placebo-Controlled Trial Examining the Effects of Cannabigerol on Indicators of Attention-Deficit/Hyperactivity Disorder
Brief Title: The Effects of Cannabigerol on Attention-Deficit/Hyperactivity Disorder
Acronym: CBG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Ellen Leen-Feldner, Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2309494774
Record Dates: First submitted 2023-10-10; First posted 2023-11-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — cannabigerol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and researchers interacting with participants will be blind to condition. An unblinded researcher team will randomize and label all pipettes containing CBG or placebo prior to each participants' session. Participants will receive individual, 1 mL pipettes containing CBG and placebo (pipettes are indistinguishable).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabigerol (Active Comparator): 1mL of 80mg of Cannabigerol. Cannabigerol is a safe, legal, non-high-inducing cannabinoid obtained from the cannabis plant.
  Interventions: Drug: Cannabigerol
- Placebo (Placebo Comparator): 1mL of Placebo. Placebo is made in the form of MCT oil.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cannabigerol — 1 mL of 80mg Cannabigerol once during experimental session
  Arms: Cannabigerol
Other: Placebo — 1 mL of placebo once during experimental session
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the effects of Cannabigerol (CBG) on indicators of Attention-Deficit/Hyperactivity Disorder (ADHD) in a sample of participants indicating/reporting symptoms associated with ADHD. The main question it aims to answer is: Does CBG reduce ADHD-related indicators relative to placebo? Participants will administer an acute dose of placebo or 80mg CBG and complete outcome measures at 45 minutes and 75 minutes. Daily surveys to monitor safety will be administered for one week following administration.

ELIGIBILITY:
1. Between 18 and 55-years-old.
2. BMI between 18 and 35 kg/m2.
3. Score a 4 or above on the Adult ADHD Self-Report Scale (ASRS-v1.1) Symptom Checklist Part A.
4. Meet diagnostic criteria for ADHD with a current severity rating of at least mild as defined by the DIAMOND.
5. Are not pregnant or currently breastfeeding.
6. Have no history of significant allergic condition, hypersensitivity, or allergic reactions to cannabis, cannabinoid medications, hemp products, medium chain triglyceride oil, or peppermint.
7. Have not used CBG or any other cannabinoid products in the past 30 days.
8. Willing to abstain from using cannabis or any THC-containing product for the duration of the study.
9. Have never used a synthetic cannabinoid or cannabinoid analogue (e.g., dronabinol, nabilone), or a synthetic cannabinoid receptor agonist (e.g., spice, k2).
10. Have not been exposed to any investigational drug or device 30 days prior to screening and you have no plans to take an investigational drug during the study.
11. Willing to maintain a stable treatment regimen (i.e., no change in current medication use) for the duration of the study.
12. Not currently taking a prescription medication for ADHD and have not been prescribed a medication for ADHD in the past six months.
13. Not currently having thoughts of committing suicide
14. Does not meet criteria for current severe major depressive disorder or a substance use disorder.
15. Have not been diagnosed with bipolar disorder or psychosis.
16. Do not have an acute illness, such as a respiratory infection or other illness that would interfere with study participation; not currently taking medication for an acute illness (e.g., antibiotic).
17. Do not have history of diagnosis related to liver function and/or significantly impaired liver function (e.g., cirrhosis of the liver, hepatitis).
18. Willing to ensure they have used effective contraception (for example, oral contraception, double barrier, intra-uterine device) for 30 prior to the study and for 30 days after study completion.
19. Have access to a ride to the University of Arkansas campus for research appointments.
20. Willing to comply with current university mandates as they pertain to COVID-19 protocols (e.g., mask wearing).
21. Do not have any serious or unstable physical health conditions including neurological or renal illness.
22. Do not have any current or historical cardiovascular conditions, including hypotension, bradycardia, or heart block.
23. No atrial fibrillation, bradycardia, or tachycardia detected via mobile electrocardiogram during the in-laboratory visit.
24. No recent illicit drug use other than cannabis, or alcohol use in the 12 hours preceding the in-laboratory visit.
25. Not currently prescribed or taking the following medications:

    * Warfarin
    * Clobazam
    * Valproic acid
    * Phenobarbital
    * Mechanistic Target of Rapamycin [mTOR] Inhibitors
    * Oral tacrolimus
    * St. John's wort
    * Epidiolex
    * Escitalopram
    * Cardiovascular medications
    * Strong CYP3A4 inhibitors (e.g., ketoconazole)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-12-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sustained Attention to Response Task | 75 minutes post CBG/placebo administration
  A computerized task that measures response inhibition.
Trail Making Test-Parts A and B (TMT-A&B) | 75 minutes post CBG/placebo administration
  A paper-and-pencil task that measures
Digit Symbol Substitution Test (DSST) | 75 minutes post CBG/placebo administration
  A paper-and-pencil task that measures attention/processing speed.
Rey Auditory Verbal Learning Test (AVLT) | 75 minutes post CBG/placebo administration
  A paper-and-pencil/verbal test that measures verbal memory.
Iowa Gambling Task (IGT) | 75 minutes post CBG/placebo administration
  A computerized task that measures decision making (an indicator of impulsivity/hyperactivity).

SECONDARY OUTCOMES:
Positive and Negative Affect Scale-Expanded Version | Baseline, 45 minutes post CBG/placebo administration, 75 minutes post CBG/placebo administration
  Self-report measure of positive and negative affect. Scores range from 30-150 on each of the two types of affects, with higher scores representing greater affect.
Karolinska Sleepiness Scale | Pre CBG/placebo administration, 75 minutes post CBG/placebo administration
  Self-report measure of subjective level of sleepiness at a particular time during the day. Scores range from 1-10, with higher scores representing greater sleepiness.
Brief Irritability Test | Pre CBG/placebo administration, 75 minutes post CBG/placebo administration
  Self-report measure of irritability. Scores range from 5-30, with higher scores representing greater irritability.
Numeric Rating Scale (pain) | Pre CBG/placebo administration, 75 minutes post CBG/placebo administration
  Self-report measure of subjective level of pain. Scores range from 0-10, with higher scores representing greater pain.
State-Trait Anxiety Inventory (State Version) | Pre CBG/placebo administration, 75 minutes post CBG/placebo administration
  Self-report measure of state anxiety. Scores range from 20 to 80 with higher scores indicating greater anxiety.
Visual Analog Scales | 75 minutes post CBG/placebo administration
  Self-report of state-like states (e.g., anxiety, hunger). This scale ranges from 0 to 100 with higher scores indicating higher levels of the indication.
Global Impression of Change | 75 minutes post CBG/placebo administration
  Self-report measure of perceived change in ADHD symptoms. This scale ranges from 1 to 7 with higher scores indicating greater improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W Leen-Feldner, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual participant data (including data dictionaries) that underlie results reported in each published report will be shared (text, tables, figures, appendices)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9months and ending 36 months following publication
Access Criteria: Researchers who provide a methodologically sound proposal. Inquiries should be directed to eleenfe@uark.edu; Requestors will need to sign a data agreement to gain access